CLINICAL TRIAL: NCT05855551
Title: Joint Interventions to Improve Birth Outcomes and Nutrition in Bangladesh: the Jibon Trial
Brief Title: Improving Birth Outcomes in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHND-Jibon
Record Dates: First submitted 2020-02-16; First posted 2023-05-11 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Birth Weight; Small for Gestational Age at Delivery; Diet; Deficiency; Gestational Weight Gain
MeSH Terms: conditions — Birth Weight; Malnutrition; Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - base cash + BCC (Experimental): pregnant women in this arm will receive the standard package (800 BDT each month), and in addition intensive group-based BCC on nutrition with a focus on how to improve their dietary intake during pregnancy
  Interventions: Other: Base cash transfer; Behavioral: Behavior change communication (BCC)
- Arm 2 - base cash + BCC + food (Experimental): pregnant women in this arm will receive the standard package (i.e., arm 1) and in addition a monthly food basket. The monthly food basket will provide 10 kg micronutrient fortified rice, 3.5 kg of lentils, and 1000 ml of oil, valued at 1000 BDT.
  Interventions: Other: Base cash transfer; Behavioral: Behavior change communication (BCC); Other: Food basket
- Arm 3 - base cash + BCC + top-up cash (Experimental): pregnant women in this arm will receive the standard package (i.e., arm 1) and in addition a monthly top-up cash of 1000 BDT to be added to the "base" amount that is part of the standard program.
  Interventions: Other: Base cash transfer; Behavioral: Behavior change communication (BCC); Other: Top-up cash

INTERVENTIONS:
Other: Base cash transfer — Program beneficiaries will receive a monthly transfer of 800 BDT. A government-to-person (G2P) payment system will be used, which will transfer cash on a monthly basis. Under this new system, beneficiaries will select one of the following payment channels based on convenience: mobile financial services or through a bank transfer (which women in remote areas could access through agent banking). Each month, women will receive a text message from the government informing her that the money has been credited to her account.
Behavioral: Behavior change communication (BCC) — The BCC strategy has two different components:
  * Monthly courtyard meetings: Courtyard sessions (12 to 15 women) will be organized at a place no more than 15 to 20 minutes walking distance from the beneficiary's home. Family members (husband, mother-in-law, …) are invited to join the meeting. Sessions are part of a continuous 4-session cycle. Each session will lasts 1.5 hours and will use different didactic methods. Topics include pregnancy nutrition and care, breastfeeding, importance of different micronutrients, and nutrition and care during lactation. The importance of a healthy diet during pregnancy is repeated in each session. Pregnant women receive a take-home poster that summarizes how to eat a healthy diet during pregnancy.
  * Home visits: Visits will cover the content of any sessions missed by pregnant women and will reinforce the messages regarding maternal diet on the take-home poster.
Other: Food basket — The monthly food basket will provide 10 kg micronutrient fortified rice , 3.5 kg of lentils, and 1000 ml of oil, valued at 800 BDT . Assuming a the ration is split equally among the 5 members of an average-sized household in rural Bangladesh and using food composition data for Bangladesh, the food basket is estimated to provide 354 kcal and 11 g of protein per person per day. The food basket will be provided once every month.
  The individually packaged foods will be distributed at the Union parishad office, community clinic, or another government facility in the first week of each month. The UDW will inform the beneficiaries of the place and time of the food distribution. Recipients will only receive the food when they present their food card. The card will also be used to record receipt of each ration. If beneficiaries cannot attend the food distribution themselves, a designated "nominee" can pick up the ration on their behalf.
  Arms: Arm 2 - base cash + BCC + food
Other: Top-up cash — The monthly top-up cash of 1,000 BDT will be added to the "base" amount that is part of the standard program. For the top-up cash transfer, a person-to-person payment system is used. WFP will contract with one popular mobile banking service (either bKash or Rockets) for the monthly top-up cash transfers. About two weeks after receiving the base cash transfer, women will receive the top-up cash through a mobile account (which can also be used to receive the base cash transfer). A text message will be sent to the beneficiary to inform her that the top-up transfer has been made into her account.
  Arms: Arm 3 - base cash + BCC + top-up cash

SUMMARY:
Maternal undernutrition is a global public health problem with far-reaching effects for both mothers and infants. Poor maternal nutrition negatively affects fetal growth and development. Both micro and macro-nutrients are required for the physiological changes and increased metabolic demands during pregnancy, including fetal growth and development. Women in Bangladesh have poor diets and are struggling to meet their nutrient requirements, especially during pregnancy and lactation when requirements are higher. Maternal undernutrition during pregnancy is associated with a range of adverse birth outcomes, including stillbirths, preterm births, low birthweight, and small-for-gestational-age (SGA) neonates, all of which remain unacceptably high in Bangladesh.

Social protection provides a promising platform on which to leverage improvements in nutrition at scale, but current evidence on the impacts of social protection on birth outcomes is limited: few studies have been conducted and some of these studies suffer from methodological limitations. The planned study will contribute to filling this knowledge gap. An additional motivation for the study is provided by the recent WHO 2016 Antenatal Care Guidelines. The guidelines call for studies on the effectiveness of alternatives to providing energy and protein supplements to pregnant women (which is recommended in undernourished populations). Studying the effectiveness of providing combinations of food and cash will help build this evidence base. A third reason to conduct the study is that both food transfers and cash transfers are commonly used policy instruments in Bangladesh, and the choice of intervention components to scale up in the CBP will be guided by the findings from this pilot study. The study findings will thus be highly policy relevant.

A three-arm cluster-randomized, non-masked, community-based, longitudinal trial will be used. Groups of pregnant women will be randomly assigned to one of three study arms providing different combinations of cash and food transfers.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with their first or second child (in case of death of the first or second child during pregnancy or within two years of birth, the mother will be eligible during her third pregnancy);
* In possession of a valid NID (or a NID application acknowledgement).
* Meeting the eligibility criteria of the Government of Bangladesh' Mother and Child Benefit Programme (MCBP)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4620 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Gestational weekly weight gain 2nd to 3rd trimester | Third pregnancy trimester (34 ± 1 wk of pregnancy)
  Women's weekly weight gain will be calculated by differencing women's weight obtained in the second and third trimester and dividing by the number of weeks between both measurements.
Total gestational weight gain by the third trimester | Third pregnancy trimester (34 ± 1 wk of pregnancy)
  Total weight gain will be calculated by calculating the difference between women's third trimester weight and the weight obtained at the time of the census.
Dietary energy intake and proportion of women below 85% of the estimate energy requirement (EER) | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  Dietary energy intake will be assessed using a 24-hour recall in the second and third trimester (18). EER will be calculated using each woman's basal metabolic rate (estimated from the woman's age, gender, and current weight), level of physical activity, and pregnancy trimester. Factors of 1.4 for low, 1.7 for moderate, and 2.0 for high physical activity will be used (19). Additional energy requirement for the second and third trimester of pregnancy (340-350 kcal/d and 452-500 kcal/d, respectively, depending on which reference will be used (20,21)) will be added to account for gestational weight gain and increases in basal metabolic rate.
Dietary protein intake | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  The 24-hour recall data will be used to assess women's protein intake.
Mean probability of micronutrient adequacy | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  the mean of the probabilities of adequacy for 11 key micronutrients (iron, calcium, zinc, vitamin A, thiamin, riboflavin, niacin, vitamin B-6, vitamin B-12, vitamin C, and folate) will be calculated using the 24h recall data. The estimated usual intake will be used to calculate the probability that the usual intake was above the EAR during pregnancy (25).
Length of gestation | Delivery
  The difference between the date of birth and the first day of the last menstrual period (assessed in the first survey) will be used to calculate length of gestation.
Preterm birth | Delivery
  Using the length of gestation, we will determine the proportion of children born before 37 weeks of gestation.
Prevalence of emotional violence towards the pregnant woman/mother of the newborn child | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Prevalence of any emotional intimate partner violence in the past 6 months measured using the WHO Violence Against Women instrument (26)
Prevalence of controlling behaviors towards the pregnant woman/mother of the newborn child | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Prevalence of any controlling behaviors in the past 6 months measured using the WHO Violence Against Women instrument (26).
Prevalence of physical violence towards the pregnant woman/mother of the newborn child | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Prevalence of any physical intimate partner violence in the past 6 months measured using the WHO Violence Against Women instrument (26)
Stress of the pregnant woman/mother of the newborn child | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Measured using women's Perceived Stress Scale score
Maternal-fetal attachment | Third pregnancy trimester (34 ± 1 wk of pregnancy)
  Maternal attachment to their unborn child will be assessed during their 3rd trimester of pregnancy using the Prenatal Attachment Inventory
Maternal-infant attachment | Two months post-partum (61 d ± 1 wk)
  Maternal attachment to their infant will be assessed at 2 months (i.e., 61 days) postpartum using the Postpartum Bonding Questionnaire
Stress of the husband of the pregnant woman | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  Measured using men's Perceived Stress Scale score (27).
Birthweight | Within 72 hours post partum
  Birthweight will be assessed within 48 to 72 hours after delivery to avoid the influence of transitory neonatal weight loss that typically happens during the first days of life.
Low birthweight | Within 72 hours post partum
  Birthweight will be assessed within 48 to 72 hours after delivery to avoid the influence of transitory neonatal weight loss that typically happens during the first days of life. Low birthweight will be defined as a weight below 2500g.
Household food security | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  The Household Food Insecurity Access Scale will be used to measure household food security status.
Value of total household consumption | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  Aggregate value of household food and non-food consumption expenditures. This is a continuous measure calculated from household survey responses on consumption behavior, using the methodology and questionnaire modules described by Deaton and Zaidi (32).
Value of household food consumption | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  Value of household food consumption expenditures. This is a continuous measure calculated from household survey responses on consumption behavior, using the methodology and questionnaire modules described by Deaton and Zaidi (32).

SECONDARY OUTCOMES:
Gestational weekly weight gain up to the 2nd trimester | Second pregnancy trimester
  Women's weekly weight gain will be calculated by differencing women's weight obtained at the census (before pregnancy) and second trimester and dividing by gestational age in weeks.
Use of iron-folic acid, calcium, vitamin B complex, and multiple micronutrient supplements | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  Women will be asked to report on their use of these supplements during pregnancy.
Antenatal care utilization by the pregnant woman | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  Antenatal care utilization will be assessed with respect to current recommendations in Bangladesh and with respect to the new WHO guidelines
Prenatal nutrition knowledge of the pregnant woman | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  Women's knowledge related to nutrition will be assessed using a set of questions developed for this study.
Post natal care utilization by the mother of the newborn child | Two months post-partum (61 d ± 1 wk)
  Postnatal care utilization will be assessed
Postpartum weight | Two months post-partum (61 d ± 1 wk)
  We will measure women's weight at the 2-month postpartum visit.
Spousal relationship between the pregnant woman/mother of the newborn child and her husband | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Measured using women's spousal relationship modules developed for the survey.
Decisionmaking by the pregnant woman/mother of the newborn child | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Measured using women's decision-making modules adapted from pro-WEAI (34).
Mobility of the pregnant woman | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Measured using mobility modules adapted from pro-WEAI (34).
Labor force participation of the pregnant woman | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  Measured using women's labor modules developed for the survey.
Attitudes toward gender and intimate partner violence of the pregnant woman | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Measured using women's attitudes toward gender and intimate partner violence modules developed for the survey.
Social capital of the pregnant woman | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Measured using modules on women's social interactions and perceptions of neighborhood responses to intimate partner violence, developed for the survey.
Agency of the pregnant woman | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Measured using women's responses on locus of control (35).
Prevalence of individual acts of intimate partner violence towards the pregnant woman/mother of the newborn child | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Prevalence of individual acts of intimate partner violence in the past 6 months measured using the WHO Violence Against Women instrument (26)
Institutional delivery | Within 72 hours post partum
  We will ask if the baby was delivered in a health facility
Skilled attendance at birth | Within 72 hours post partum
  Women will be asked if a skilled birth attended the birth of the child
Caesarian section | Within 72 hours post partum
  Women will be asked if a c-section was used to deliver the child
Prenatal nutrition knowledge of the husband of the pregnant woman | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  Using a similar approach as that use for pregnant women, husband's nutrition knowledge.
Husband's weight | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  Weight of the husband will be assessed.
Birth length | Within 72 hours post partum
  The length of the newborn will be assessed at the time of the birthweight assessment.
Infant length and weight | Two months post-partum (61 d ± 1 wk)
  Length and weight at 2 mo postpartum
Colostrum intake, time between birth and putting infant to breast, (exclusive) breastfeeding after birth | Within 72 hours post partum
  Women will be asked whether and how they breastfeed their newborn child. We will also assess if other liquids are provided to the child (36).
(Exclusive) breastfeeding and infant feeding practices at 2 months | Two months post-partum (61 d ± 1 wk)
  women will be asked whether and how they breastfeed their newborn child. We will also assess if other liquids and solid foods are provided to the child (36).
Neonatal and infant mortality | One and two months post-partum
  neonatal (within the first 1 month after birth) and infant (within the first 2 months after birth) mortality will be assessed through parental recall at the 2-month postpartum visit.
Value of household non-food consumption | Second and third pregnancy trimester (34 ± 1 wk of pregnancy)
  Value of household non-food consumption expenditures. This is a continuous measure calculated from household survey responses on consumption behavior, using the methodology and questionnaire modules described by Deaton and Zaidi (32). The third-trimester assessment will be used to assess impact.
Housing quality | Second pregnancy trimester; Two months post-partum (61 d ± 1 wk)
  Quality of housing stock, measured using a module developed for the study context and collected through household enumerator observation during interviews.
Household asset ownership | Second pregnancy trimester; Two months post-partum (61 d ± 1 wk)
  Index of household asset ownership, measured using a module developed for the study context.
Household income from remittances | Third pregnancy trimester (34 ± 1 wk of pregnancy)
  Measured with a module on income (Taka) from remittances received from relatives outside and within the country. The third-trimester assessment will be used to assess impact
Household savings | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  A continuous measure on total household savings, calculated using reported savings of each household member 15 years of age or older.
Household loans | Second and third pregnancy trimester (34 ± 1 wk of pregnancy); Two months post-partum (61 d ± 1 wk)
  A continuous measure on household loans, calculated using reported amounts of loans taken and outstanding amounts owed for each household member 15 years of age or older.

OTHER OUTCOMES:
Program enrollment | Second and third pregnancy trimester (34 ± 1 wk of pregnancy), 2 months postpartum
  enrollment in the MCBP program
Receipt of program benefits (base cash, food, top-up cash) and participation in BCC sessions | Second and third pregnancy trimester (34 ± 1 wk of pregnancy), 2 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Jef Leroy, PhD, Principal Investigator — International Food Policy Research Institute; Shalini Roy, PhD, Principal Investigator — International Food Policy Research Institute
Locations (1):
- rural areas in 6 upazilas in Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of primary data analyses

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT05855551/SAP_000.pdf